CLINICAL TRIAL: NCT06102369
Title: The Role of Narrow Band Imaging (NBI) Bronchoscopy in Detecting Bronchial Squamous Dysplasia in Lung Cancer
Status: Enrolling by invitation | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Mia Elhidsi, MD, Principal Investigator, Fakultas Kedokteran Universitas Indonesia
Other Study IDs: ND-552/UN2.RST/PPM.00.00/2023
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Pulmonary Cancer; Lung Cancer
Keywords: bronchoscopy; narrow-band imaging (NBI); lung cancer; bronchial squamous dysplasia
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — formalin-fixed paraffin-embedded (FFPE) tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigators conducted an observational diagnostic study. The primary objective of the study is to develop a scoring system for detecting pre-lung cancer abnormalities using narrow-band imaging (NBI) bronchoscopy. From the collected data, investigators will perform a multivariate analysis based on the odds ratio (OR) using IBM SPSS software. The result of the data analysis will be transformed into a scoring system aimed to facilitate the early diagnosis of lung cancer, specifically at the pre-cancer stage. This scoring system will also help clinicians detect pre-cancerous abnormalities early and improve patient recovery prospects.

Several research questions to be addressed are as follows:

1. What are the NBI image criteria for detecting pre-cancerous lesions in lung tumor patients?
2. What is the diagnostic profile of NBI bronchoscopy in detecting pre-cancerous lesions in lung tumor patients?
3. Can adding the NBI bronchoscopy procedure to the standard bronchoscopy procedure enhance the diagnostic accuracy in detecting pre-cancerous lesions in lung tumor patients?

The study population consists of lung tumor patients who have undergone bronchoscopy procedures and meet the protocol acceptance criteria. Bronchial biopsies will be collected from these patients, followed by histopathological examinations.

DETAILED DESCRIPTION:
1. Study Design: This is an observational diagnostic study. The research was conducted at the Central Surgical Installation (CSI) of Persahabatan Hospital, where bronchoscopy procedures, bronchial biopsy collection, and specimen handling took place. The histopathological examinations were carried out in the Department of Anatomical Pathology, Faculty of Medicine, Universitas Indonesia, Cipto Mangunkusumo National General Hospital. The patient recruitment time ranges from March to December 2023.
2. Population: The target population consists of all lung tumor patients. The accessible population consisted of lung tumor patients who underwent bronchoscopy procedures at Persahabatan Hospital from March to December 2023.
3. The study participants: The study participants comprised individuals from the accessible population who met the research subject acceptance criteria and provided informed consent. The consecutive sampling method was employed.
4. Study participants size calculation: The study participants size was calculated using the diagnostic research sample size formula. The minimum study participants size required was 110 subjects.
5. Inclusion criteria:

   * Patient aged > 18 years undergoing bronchoscopy for diagnostic evaluation of lung tumors
   * Recent radiological examinations, including both chest X-ray and chest CT scans, within the last month, revealed a central lesion of lung cancer
6. Exclusion criteria:

   * Refusal to provide informed consent
   * Contraindications to bronchoscopy
7. Study participants selection: Screening was conducted on all lung tumor patients scheduled for bronchoscopy procedures, and the study participants selection was carried out in accordance with the inclusion and exclusion criteria
8. Sampling Technique:

   The preparation and execution of bronchoscopy and bronchial biopsy were performed in accordance with the standard operating procedures (SOP) at Persahabatan Hospital. The bronchoscopy and bronchial biopsy procedures were conducted by a single operator, the principal investigator. The bronchoscopy procedure uses general anesthesia. The flexible fiberoptic bronchoscopy was performed using an Olympus EVIS EXERA III with a Xenon light source, model CLV-190, and BF-1TQ170 series scope. The Boston Scientific Radial JawTM 4 disposable lung biopsy forceps were employed. Bronchoscopy was initially conducted under the white light, followed by narrow-spectrum light. The NBI assessment was performed in two areas, consisting of area 1 (trachea and carina) and area 2 (right main bronchus, right upper lobe orifice, truncus intermedius, right lower lobe orifice, left main bronchus, left upper lobe orifice, and left lower lobe orifice). Biopsies were taken from both areas based on the NBI bronchoscopy findings. Tissue from each area was placed in a separate 10% formalin solution. Tissue processing involved paraffin embedding and Hematoxylin-Eosin staining. Tissue processing was performed using a Tissue Processor machine. Following tissue processing, paraffin blocks were created and sectioned. Hematoxylin-Eosin staining was then performed. Diagnosis of squamous bronchial dysplasia (pre-cancer lesion) was made by a specialist in Anatomical Pathology.
9. Data analysis: The research data were recorded on research forms and subsequently entered into SPSS 26 software. the bivariate analysis was conducted between each vascular pattern based on NBI bronchoscopy and the histopathological result. The descriptive data will be presented by the text and tables consist of the basic characteristics of the study participants and research variables. The multivariate analysis was performed on all vascular patterns based on NBI bronchoscopy and histopathological results. Furthermore, a pre-cancer prediction score was generated. An analysis of the AUC (area under the curve) of the squamous dysplasia prediction model form NBI bronchoscopy findings was conducted with a significance level set at p < 0.0.5

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years undergoing bronchoscopy for diagnostic evaluation of lung tumors.
* Recent radiological examinations, including both chest X-rays and chest CT scans, within the last month, revealed central lesions.

Exclusion Criteria:

* Refusal to provide informed consent
* Contraindications to bronchoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Population: The target population consists of all lung tumor patients. The accessible population consisted of lung tumor patients who underwent bronchoscopy procedures at Persahabatan Hospital from March to December 2023.
  2. The study participants: The study participants comprised individuals from the accessible population who met the research subject acceptance criteria and provided informed consent. The consecutive sampling method was employed.
  3. The study participants size calculation: The study participants size was calculated using the diagnostic research sample size formula. The minimum study participants size required was 110 subjects.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
To determine the sensitivity, specificity, positive predictive value, and negative predictive value of the bronchoscopic narrow-band imaging (NBI) in detecting bronchial squamous dysplasia | Based on the research timeline, all statistical analysis and data processing will be conducted from January to February 2024
  To address this outome, researchers will utilize parameters derived form NBI bronchoscopy images, consist of normal vascularity, increased vascular frequency, dotted, spiral, tortuous and abrupt-ending blood vessels (on a nominal scale). These parameters will be employed in conjunction with histopathological images (dysplasia or non dysplasia) for comparative analysis

SECONDARY OUTCOMES:
To determine the proportion of bronchial squamous dysplasia in lung cancer patients | Based on the research timeline, all statistical analysis and data processing will be conducted from January to February 2024
  This refers to the ratio of the number of cases with squamous bronchial dysplasia to the total number of lung cancer patients in the study. The proportion measures how much squamous bronchial dysplasia is found in lung cancer patients within the study population (descriptive analysis)
To establish the correlation between the NBI bronchoscopy findings and bronchial squamous dysplasia in lung cancer patients | Based on the research timeline, all statistical analysis and data processing will be conducted from January to February 2024
  Researchers will utilize parameters derived form NBI bronchoscopy images, consist of normal vascularity, increased vascular frequency, dotted, spiral, tortuous and abrupt-ending blood vessels (on a nominal scale). These parameters will be employed in conjunction with histopathological images (dysplasia or non dysplasia). Additionally, bivariate analysis followed by multivariate logistic regression analysis is conducted between the NBI bronchoscopy image and squamous bronchial dysplasia.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
Researchers might be engaging in consultations with ethics boards, legal experts, and stakeholders to develop a robust and ethical sharing plan that adheres to the highest standards of privacy and security.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT06102369/Prot_SAP_ICF_001.pdf